CLINICAL TRIAL: NCT06306872
Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ABSK061 Minitablets Following Single and Multiple Oral Doses and to Assess the Effect of Administration With Soft Foods in Healthy Adults
Brief Title: A Clinical Trial to Evaluate the Relative Bioavailability of New and Old ABSK-011 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ABSK-011-102
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 1:1 to arms A (Sequence A) or arms B (Sequence B) to receive a single dose of ABSK-011 orally in two separate doses, spaced at least 4 days apart. Among them, subjects in sequence A will be given ABSK-011 220 mg (100 mg capsule *2 and 20 mg capsule *1) and ABSK-011 200 mg (100 mg capsule *2) on an empty stomach in the morning of the first day of cycle 1 (C1D1) and the first day of cycle 2 (C2D1), respectively. Subjects in sequence B will be given ABSK-011 new formulation 200 mg (100 mg capsule *2) and ABSK-011 old formulation 220 mg (100 mg capsule *2 and 20 mg capsule *1) on an empty stomach in the morning of Cycle 1 day (C1D1) and cycle 2 day (C2D1), respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Other): Subjects in sequence A will be given ABSK-011 old formulation 220 mg (100 mg capsule *2 and 20 mg capsule *1) on an empty stomach in the morning of the first day of cycle 1 (C1D1) and ABSK-011 new formulation 200 mg (100 mg capsule *2) on an empty stomach in the morning of the first day of cycle 2 (C2D1).
  Interventions: Drug: Sequence A ABSK-011
- Sequence B (Other): Subjects in sequence B will be given ABSK-011 new formulation 200 mg (100 mg capsule *2) on an empty stomach in the morning of Cycle 1 day (C1D1) and ABSK-011 old formulation 220 mg (100 mg capsule *2 and 20 mg capsule *1) on an empty stomach in the morning of the first day of cycle 2 (C2D1).
  Interventions: Drug: Sequence B ABSK-011

INTERVENTIONS:
Drug: Sequence A ABSK-011 — Subjects in sequence A will receive 220 mg (100 mg capsule *2 and 20 mg capsule *1) Oral administration of ABSK-011 old formulation at the first day of cycle 1 (C1D1), followed by a washout period of at least 4 days.Subjects will receive 200 mg(100 mg capsule *2) Oral administration of ABSK-011 new formulation at the first day of cycle 2 (C2D1).
  Arms: Sequence A
Drug: Sequence B ABSK-011 — Subjects in sequence A will receive 200 mg(100 mg capsule *2) Oral administration of ABSK-011 old formulation at the first day of cycle 1 (C1D1), followed by a washout period of at least 4 days.Subjects will receive 220 mg (100 mg capsule *2 and 20 mg capsule *1) Oral administration of ABSK-011 new formulation at the first day of cycle 2 (C2D1).
  Arms: Sequence B

SUMMARY:
The main objective of which is to evaluate the relative bioavailability and PK characteristics of new and old ABSK-011 capsules in a single oral dose

DETAILED DESCRIPTION:
This study consists of three separate parts: Part A, Part B and Part C. Part A is designed as a two-period, open-label, two-sequence crossover study, the main objective of which is to evaluate the relative bioavailability and PK characteristics of new and old ABSK-011 capsules in a single oral dose.

Part B is designed as a three-period, open-label, three-sequence crossover study, the main objective of which is to evaluate the relative bioavailability and PK characteristics of new ABSK-011 formulation versus the old formulation at high and low doses for single oral administration.

Part C was designed as a four-period, open-label, fixed-sequence study, the main objective of which was to evaluate the effects of low-fat diet, high-fat diet and omeprazole magnesium enteric-coated tablets on PK of the new ABSK-011 formulation after a single oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged between 18 and 45 years (including 18 and 45 years) at the time of screening;
2. Male ≥50 kg, female ≥45kg, body mass index (BMI) between 19 and 28 (including 19 and 28), BMI= weight (kg)/height (m) 2;
3. Physical examination, laboratory examination and other relevant examination results before the first medication are normal or abnormal but meet the following requirements, or other abnormal results but not clinically significant determined by the investigator:

   1. 35.9℃≤ ear temperature ≤37.5℃;
   2. pulse rate ≥55 times/min and ≤100 times/min;
   3. Systolic blood pressure ≥90 mmHg and < 140 mmHg, diastolic blood pressure ≥60mmHg and < 90 mmHg;
   4. Total bilirubin (TBIL) ≤1.5×ULN;
4. Fertile male or female subjects must consent to the use of an effective contraceptive method during the study period and for 6 months after the last dose of the investigational drug is administered (And male subjects do not donate sperm during this period, and female subjects do not donate eggs during this period; Female subjects must be non-pregnant and non-lactating female subjects, defined as women in a state of pregnancy from conception to termination of pregnancy, as determined by laboratory human chorionic gonadotropin (hCG) test within 7 days before the start of the study;
5. Voluntarily participate in this clinical trial, understand the study procedure and sign the informed consent before screening; Good compliance, willing to follow study procedures.

Exclusion Criteria:

1. Patients with medical history or existing diseases of motor system, neuropsychiatric system, endocrine system, blood circulatory system, respiratory system, digestive system, urinary system, reproductive system, and other abnormalities, and those determined by the investigator to be clinically significant ;
2. A known or persistent mental disorder that may interfere with the participant's participation in the study, as determined by the investigator;
3. Known allergic history to food, environment, experimental drug ABSK-011 or other drugs;
4. Participants who have participated in other clinical trials and used other clinical trial drugs or test devices within 3 months before or during the screening period, or plan to participate in other clinical trials during the study period, or participants who do not participate in clinical trials themselves;\
5. have previously participated in this study or any other study related to ABSK-011 as a subject and have taken ABSK-011;
6. Patients who had used proton pump inhibitors (including omeprazole, Lansoprazole, Rabeprazole, pantoprazole, etc.) within 14 days before the first dose;
7. Those who have used strong inhibitors or inducers of CYP3A4 (including grapefruit juice, grapefruit hybrids, pomegranates, star fruits, grapefruits, Seville oranges and fruit juices or other processed products) within 14 days before the first dose, or have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products;
8. For those who have used CYP2C19 inhibitors or inducers (including fluoxetine, fluvoxamine, ticlopidine, rifamepine) within 14 days before the first dose, (Part C only);
9. There are factors that significantly affect drug absorption, distribution, metabolism and excretion, such as inability to take oral experimental drugs (dysphagia), significant nausea, vomiting and malabsorption, history of gastric or intestinal surgery, or other surgical history that affects drug absorption, distribution, metabolism and excretion (except appendicitis surgery);
10. Patients with needle fainting, blood fainting history, or inability to tolerate venipunction, or difficulty in blood collection;
11. Blood donation or heavy blood loss (≥400ml) within 3 months before or during screening (except female menstrual period);
12. Have special dietary requirements, can not comply with the unified diet (such as the standard meal food intolerance, lactose intolerance, etc.) and the corresponding regulations, or have swallowing difficulties;
13. Those who do not wish to comply with the dietary requirements/restrictions during the study period, which are: (i) only dietary supplements provided by the study center during hospitalization, (ii) avoiding CYP3A4 strong inhibitor or inducer during the study, and (iii) avoiding other CYP2C19 strong inhibitor or inducer during the study ( (iii) Only Part C);
14. Those who consumed more than 14 units of alcohol per week in the 3 months prior to screening (1 unit of alcohol is about 360mL beer or 45mL spirits with 40% alcohol or 150mL wine), or whose alcohol breath test results were > 0mg/100ml, or those who cannot abstain from alcohol during the study;
15. Smokers who smoked more than 5 cigarettes per day (or a corresponding amount of tobacco or nicotine products) in the 3 months prior to screening; Or unable to stop using any tobacco products during the trial;
16. People who had excessive methylxanthine/caffeine consumption in the past 6 months (excess consumption was defined as consuming more than 6 units of caffeine per day, with 1 unit of caffeine equivalent to 177 ml of coffee, 355 ml of tea, 355 ml of cola, or 85 grams of chocolate), Or were unwilling to comply with the methylxanthine/caffeine use restrictions in 5.3.3 during the study period, or had a known history of substance abuse or screened positive for substance abuse;
17. Hepatitis B surface antigen, treponema pallidum antibody, antibody to human immunodeficiency virus, antibody to hepatitis C antibody were abnormal and were clinically significant determined by the investigator;
18. Patients with a history of bacterial, fungal, parasitic, viral (excluding nasopharyngitis) or mycobacterium infection within 45 days prior to the first administration, or imaging findings (chest radiograph) supporting related infections (as determined by the investigator);
19. had been vaccinated within 2 months prior to the first dose, or intended to be vaccinated throughout the study period;
20. Any other factors that the investigator considers inappropriate for participation in this trial, which may affect the participant's adherence to the protocol, interfere with the interpretation of the study results, or expose the participant to risk. Or subjects withdraw from the experiment for their own reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Cmax | From pre-dose up to 72 hours post-dose. assessed up to 12 months
  Maximum observed concentration
AUC | From pre-dose up to 72 hours post-dose. assessed up to 12 months
  Area under the concentration-time curve
tmax | From pre-dose up to 72 hours post-dose. assessed up to 12 months
  Time to maximum observed concentration

SECONDARY OUTCOMES:
AEs | The date of signing the informed consent form until 30 days (including Day 30) after the last dose of study drug, assessed up to 12 months.
  Adverse events
SAEs SAEs | The date of signing the informed consent form until 30 days (including Day 30) after the last dose of study drug, assessed up to 12 months.
  Serious adverse events (SAEs)
t1/2 | From pre-dose up to 72 hours post-dose. assessed up to 12 months
  Elimination half-life
Vz/F | From pre-dose up to 72 hours post-dose. assessed up to 12 months
  Apparent volume of distribution
CL/F CL/F | From pre-dose up to 72 hours post-dose. assessed up to 12 months
  Apparent oral clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China